CLINICAL TRIAL: NCT03712813
Title: Effect of Low Intensity Vibration (LIV) on Aromatase Inhibitor- Induced Musculoskeletal Dysfunction in Early Stage Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Tarah J Ballinger, MD, Assistant Professor of Clinical Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IUSCC-0680
Record Dates: First submitted 2018-10-16; First posted 2018-10-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: aromatase inhibitors; low intensity vibration
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio to LIV or the standard of care. The total patient enrollment will be 72 patients with 36 patients in each arm. Upon registration, subjects will be randomized and given an automated sequence number.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Macrodyne LivMD plate (Experimental)
  Interventions: Device: Macrodyne LivMD plate
- Wait-Listed Control (No Intervention)

INTERVENTIONS:
Device: Macrodyne LivMD plate — Synchronous (applied to both feet) low intensity vibration for 10 minutes, twice daily for 12 months.
  Arms: Macrodyne LivMD plate

SUMMARY:
The purpose of this study is to compare the effect of low intensity vibration (LIV) delivered for 10 minutes twice daily for 12 months on skeletal muscle function, in terms of energetic capacity measured by power generation on a stationary bicycle, among patients with early stage breast cancer planned to initiate aromatase inhibitor therapy who do not currently participate in regular exercise, compared to a wait- listed control.

DETAILED DESCRIPTION:
This is a randomized phase II, two arm, single-center study designed to compare the effect of LIV versus wait-list control on the clinical parameter of energetic capacity, or power generation, in patients with early stage breast cancer receiving aromatase inhibitor therapy over a 12-month period. The primary endpoint is the 12-month change in energetic capacity since baseline.

Primary Objective To compare the effect of LIV delivered for 10 minutes twice daily for 12 months on skeletal muscle function, in terms of energetic capacity measured by power generation on a stationary bicycle, among patients with early stage breast cancer planned to initiate aromatase inhibitor therapy who do not currently participate in regular exercise, compared to a wait- listed control

Secondary Objectives

1. To compare the effect of LIV versus wait-listed control upon muscle contractile properties including peak power, fatigue resistance, and recovery, measured by isokinetic knee extension
2. To compare the effect of LIV versus wait- listed control upon body composition (lean mass, total adiposity) measured by DXA scan
3. To compare the effect of LIV versus wait- listed control upon bone mineral density (T score) measured by DXA scan
4. To compare the effect of LIV versus wait- listed control upon muscle adipose infiltration measured by muscle density on peripheral quantitative CT imaging of the proximal and distal tibia and radius
5. To compare the effect of LIV versus wait-listed control on trabecular and cortical volumetric bone mineral density by high resolution peripheral quantitative CT of the distal and diaphyseal tibia and radius
6. To compare the effect of LIV versus wait- listed control on serologic markers of bone turnover, including TGF-beta and NTX
7. To compare the effect of LIV versus wait- listed controls upon patient reported outcome measures of fatigue (measured by the Basic Fatigue Inventory), muscle ache, and joint pain (measured by PRO-CTCAE)
8. To describe the feasibility of LIV in this patient population, defined by patient compliance and follow up with the intervention

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Diagnosis of DCIS or stage I, II, or III breast cancer 3 Planned to initiate an AI

   1. Post- menopausal defined as ≥ 60 years of age, prior bilateral oophorectomy, or age over 50 and absence of any menstrual periods in the last 12 months, or FSH and estradiol in the menopausal range
   2. Premenopausal patients receiving chemical ovarian suppression are allowed
   3. Prior aromatase inhibitor use (if this is a second primary, for example) is allowed as long as it has been more than 12 months
   4. Prior tamoxifen is allowed if switching to an aromatase inhibitor, as long as it has been 28 days between last tamoxifen dose and the baseline procedures (per the half-life of tamoxifen)

4. Completion of all primary therapy for breast cancer, including surgery, radiation, and chemotherapy. Patients must be ≥ 21 days from chemotherapy completion and ≥14 days from radiation completion. Ongoing HER2 targeted therapy with trastuzumab or pertuzumab, or TDM1 is allowed. Ongoing therapy with abemaciclib per standard of care is allowed.

5. Baseline T score > - 2.5 on DXA 6. Body weight less than 275 lbs., as dictated by the weight limit for the LIV platforms 7. ECOG performance status of 0-2 at the time of study enrollment 8. Informed consent and authorization of the release of health information must be obtained according to institutional guidelines 9. Physically able to stand unassisted for 10 minutes at a time 10. Currently not participating in regular exercise (defined as less than 90 minutes of moderate to vigorous exercise per week measured by the RPAQ questionnaire)

Exclusion Criteria:

1. Unwilling to co-enroll onto the companion FIT core study (IRB study #1707550885)
2. Diagnosis of other disorder affecting bone function or turnover, such as Paget's disease, renal osteodystrophy, parathyroid disorders, vitamin D deficiency/osteomalacia, chronic renal disease (Cr > 1.4)

   a. Vitamin D will be checked during screening. Patients with Vit D < 20 can be enrolled if supplementation is initiated per the treating physician.
3. Prior history of non-traumatic, fragility bone fracture
4. Any muscle or neuromuscular disorder affecting muscle function, such as muscular dystrophy, myositis, or amyotrophic lateral sclerosis
5. Use of bisphosphonates or denosumab within the prior 12 months
6. History of retinal detachment
7. Current or planned pacemaker
8. Current or planned cochlear implant
9. Any condition precluding power protocol participation (i.e. riding a stationary bicycle), including: NYHA class III or IV congestive heart failure, uncontrolled angina, myocardial infarction in the prior 12 months, orthopedic surgery in the previous 6 months or plans for orthopedic surgery during the study period, chronic uncontrolled pulmonary conditions such as uncontrolled asthma (symptoms > 2 days/week) or dyspnea requiring oxygen, symptomatic peripheral vascular disease, or any other comorbidity that would interfere with the ability to complete and comply with the protocol in the opinion of the investigator
10. Metastatic breast cancer

    a. History of prior treated malignancies, other than breast cancer, that are now stable, are in remission, and do not require active therapy, are acceptable.
11. Patients requiring chronic anticoagulation are excluded from participation in the optional muscle biopsy collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2025-12-18 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Mean change in energetic capacity measured by peak power generation on a stationary bicycle | Baseline, 6 months, and 12 months
  Peak power will be measured using the Power Protocol-B

SECONDARY OUTCOMES:
Change in muscle contractile properties including peak power, fatigue resistance, and time to recovery measured by isokinetic knee extension | Baseline, 6 months, and 12 months
  A Biodex 4 system will be used to measure each subject's muscle contractile properties
Change in lean body mass | Baseline, 6 months, and 12 months
  Lean mass, total adiposity measured by DXA scan
Change in bone mineral density of the lumbar spine by T score | Baseline, 6 months, and 12 months
  Bone mineral density (T score) measured by DXA scan
Change in trabecular and cortical volumetric bone mineral density | Baseline and 12 months
  By high resolution peripheral quantitative CT of the distal and diaphyseal tibia and radius
Change in serologic bone markers of bone turnover (TGF-beta and NTX) by quantitative measurements using ELISA | Baseline and 12 months
  TGF-beta and NTX by quantitative measurements using ELISA
Patient reported fatigue measured by the Basic Fatigue Inventory score | Baseline, 6 months, and 12 months
  Average of all 9 items ranging in a score of 0-10 (total possible score of 11) scores range from 1( no fatigue/does not interfere) to 10 (as bad as you can imagine/completely interferes)
Patient reported aching muscles and joint pain measured by NCI Patient Reported Outcomes-Common Terminology Criteria for Adverse Events score | Baseline, 6 months, and 12 months
  Average of 2 scale items for aching muscles and joint pain on a 5-point Likert scale (ranging in severity) with a total possible score of 5 (i.e. very severe/ almost constantly)
Feasibility of low intensity vibration defined by patient compliance | Once monthly from Baseline to 12 months
  Patients will be asked by the study nurse how they are doing with their LIV therapy

CONTACTS AND LOCATIONS:
Overall Officials: Tarah Ballinger, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana, United States